## **Statistical Analysis of Data**

NCSS (Number Cruncher Statistical System) 2007 (Kaysville, Utah, USA) was used for statistical analysis (Serial Number: N7H5-J8E5-D4G2-H5L6-W2R7). Descriptive statistical methods (mean, standard deviation, frequency, ratio) were used in the evaluation of the study data. One-way Anova Test was used for comparison of the groups with normal distribution and Kruskal Wallis test was used for comparison of the groups with normal distribution. Paired Samples t-test was used for paired comparisons of dependent variables showing normal distribution, and Wilcoxon Signed Ranks Test was used for paired comparisons of dependent variables that did not show normal distribution. Repeated Measures Test was used for the follow-up of the variables with normal distribution and Friedman Test was used for the follow-up of the variables with the normal distribution. In order to evaluate the effect size between the groups, significance was evaluated using Cohen's Effect Size at p <0.05 level.